CLINICAL TRIAL: NCT05190250
Title: Pro-inflammatory Cytokines and Implantation Process in Women With Primary Idiopathic Infertility
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Anna Horbaczewska, Principal Investigator, Jagiellonian University
Other Study IDs: K / DSC / 0042
Record Dates: First submitted 2021-07-22; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Infertility, Female; Infertility Unexplained; Inflammatory Response
Keywords: infertility; inflammation; endometrial receptivity
MeSH Terms: conditions — Infertility, Female; Infertility; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endometrial tissue - aspiration biopsy Blood sample 5ml
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group - women with idiopathic infertility: Endometrial biopsy during implantation window Blood analysis
  Interventions: Diagnostic Test: Pipelle biopsy
- Control group - women with naturally conceived offspring: Endometrial biopsy during implantation window Blood analysis
  Interventions: Diagnostic Test: Pipelle biopsy

INTERVENTIONS:
Diagnostic Test: Pipelle biopsy — Ultrasonographically confirmed implantation window. Collection of material with use of Pipelle biopsy. Collection of 5 ml venous blood.
  Other Names: Blood sampling

SUMMARY:
Infertility is a common, worldwide problem. In about 20% of couples, the causative agent of infertility cannot be identified after routine diagnostic tests. One of the causes of idiopathic infertility may be implantation disorders.

Implantation can take place at a strictly defined moment in the menstrual cycle, when the capacity of the blastocyst to implant is overlapped with readiness for its acceptance by the endometrium, the so-called endometrial receptivity.The time interval in which the endometrium exhibits this property is called the implantation window.

The acquisition of receptivity by the endometrium is reflected in cellular and structural changes.The changes taking place at the cellular and molecular levels within the endometrium are compared to processes such as wound healing and degradation of the matrix during the neoplastic process.In considering the role of local inflammation in fertility, it is essential to distinguish between acute and chronic inflammation of moderate or low intensity.The profile of the molecules seen in a given inflammation depends on the severity, duration and mechanisms involved in the inflammation process, as well as the ability of the body's immune system to respond and adapt.IL-18 is a pro-inflammatory cytokine that mediates a type 1 cellular response. In the context of fertilization, IL-18 is a bivalent cytokine. Outside of the implantation window, IL-18 acts as an IFN-gamma inducer and is seen as a detrimental factor in the implantation process. During the implantation window, IL-18 becomes one of the main factors involved in the proper preparation of the spiral arteries. Histamine meets all the criteria of an inflammatory mediator. Histamine expression is also expressed in the endometrium, where it plays the role of a paracrine messenger during embryo decision-making and implantation. Adequate glucose uptake and metabolism are essential for the proper differentiation of the uterine endometrium towards a receptive state that allows the implantation of the embryo. The best described and most abundant glucose transporter in the endometrial stroma is GLUT1. However, there are no data on the role of GLUT4 in undetermined infertility.

GLUT4 is one of the better studied transporters because of its major role in whole body glucose homeostasis and the pathogenesis of type II diabetes.

Aims:1. Analysis of the level of interleukin 18 and histamine as molecules with a postulated role in the implantation process in the receptive endometrium in women with primary infertility of unknown etiology and comparing it to the group of women with naturally conceived offspring.

2. Assessment of the correlation of the levels of interleukin 18 and histamine in the receptive endometrium and in the blood as an attempt to find a diagnostic useful marker of receptivity.

3. Analysis of GLUT4 level in the receptive endometrium between two groups.

Materials and Methods:

Patients recruited from among women hospitalized at the CMUJ Gynecological Endocrinology Clinic for hormonal diagnostics.

1. The patient's visit during the implantation window (appropriate time of the cycle determined on the basis of ultrasound ovulation monitoring)
2. Endometrial aspiration biopsy, venous blood collection (5 ml). Preparation of material.
3. Analysis of the collected material.

DETAILED DESCRIPTION:
Infertility affects approximately 8 to 12% of reproductive age couples worldwide, equivalent to more than 186 million people.

In approximately 20% of couples, the causative agent of infertility cannot be identified after routine diagnostic tests. One of the causes of idiopathic infertility may be disorders of the implantation process.

Implantation can take place at a specific point in the menstrual cycle, when the capacity of the blastocyst to implant is overlapped with readiness for its acceptance by the endometrium, the so-called endometrial receptivity.

The time interval in which the endometrium exhibits this property is called the implantation window.

The implantation window in humans is a period of 3 to 6 days, it falls on half of the secretory phase - that is, 6 to 10 days after the LH peak.

The acquisition of receptivity by the endometrium is reflected in cellular and structural changes.

The processes are hormonally controlled by estrogens and progesterone of ovarian origin. In addition, locally produced signaling molecules such as cytokines, growth factors, and lipid mediators via autocrine, paracrine and juxtacrine signaling are important.

Genetically receptive and decisive are driven by the Hoxa10 and Hoxa11 homeobox genes, whose expression is increased by the action of steroid hormones. Changes at the cellular and molecular levels within the endometrium are compared to processes such as wound healing and degradation of the matrix during the process of cancer invasion.

Among the cells of the immune system infiltrating the endometrium, mononuclear cells dominate: macrophages, lymphocytes and NK cells.

In considering the role of local inflammation in fertility, it is essential to distinguish between acute and chronic inflammation of moderate or low intensity.

In the acute phase of the inflammatory response, cells of the immune system migrate to the site of injury in a carefully planned sequence of events facilitated by soluble mediators such as cytokines, chemokines, and acute phase proteins. Depending on the severity of the injury, this acute phase may be sufficient to repair the damage and initiate healing processes.

Prolonged inflammation, as a result of prolonged exposure to stimulation or an inappropriate response against one's own tissues, can lead to a chronic phase, in which tissue damage and fibrosis can occur.

The profile of the molecules seen in a given inflammation depends on the severity, duration and mechanisms involved in the inflammation process, as well as the ability of the body's immune system to respond and adapt.

Aim of the study was to investigate whether the levels of selected inflammatory molecules - interleukin18 and histamine, differ in the population of women with undetermined infertility compared to women with naturally conceived offspring.

Materials and methods A prospective, cross-sectional study was conducted. The study design received a positive opinion of the Bioethics Committee of the Jagiellonian University No. 1072.6120.78.2017 dated June 29, 2017 The funds were obtained from the grant No. K / DSC / 00421 of the Ministry of Science and Higher Education. The study group consisted of 58 women diagnosed with primary infertility, and a control group consisted of 8 patients with naturally conceived offspring. Patients were recruited from among women hospitalized at the Gynecological Endocrinology and Gynecology Clinic, consulted at the Gynecological Endocrinology Clinic and diagnosed under the Comprehensive Reproductive Health Program in the period from November 2017 to March 2020.

The inclusion criteria for the study group were met by women of reproductive age (18-40 years old) suffering from primary infertility (unsuccessfully trying to become pregnant for more than a year), menstruating regularly, not using hormone therapy.

The exclusion criteria were: established male factor of infertility, tubal factor, endometriosis, inflammation in the pelvic area - currently and in the history, hormonal background of infertility, obesity, insulin resistance, status post at least one miscarriage and chronic autoimmune diseases.

The inclusion criteria for the control group were met by patients of reproductive age (18-40 years) with naturally conceived offspring up to three years of age, with regular menstruation. The exclusion criteria were: condition after surgery on the uterus, including curettage of the uterine cavity, endometriosis, pelvic inflammation - present and in the history, at least one miscarriage, obesity, insulin resistance, chronic autoimmune diseases, breastfeeding.

Patients from both groups recruited for the study were examined during the implantation window. The appropriate timing of the cycle was determined by ultrasound ovulation monitoring. Patients reported around day 10 of the cycle to observe the growth of the dominant follicle. The examination was repeated after 3-4 days. If the dominant follicle growth was confirmed, the patient performed a urine LH test at home 16 days before the expected onset of menstruation. Patients reported 6-8 days after the LH peak or, in case of questionable test result, in the middle of the luteal phase determined by the reported length of the menstrual cycles - 8-4 days before the day of the expected period. During the visit, an ultrasound examination was performed to confirm past ovulation (observation of the corpus luteum in an identical ovary, endometrium at least 10 mm wide).

The patients were informed about the necessity to give up intercourse in the cycle in which the study was conducted, which was confirmed in the study documentation. Patients who did not accept this requirement could not be admitted to the study. During the visit, after ovulation was confirmed, endometrial aspiration biopsy was performed using a plastic pipette with a diameter of approx. 3 mm (Pipelle Endometrial Suction Curette). If there were difficulties in penetrating the cervical canal with a pipette, the upper lip of the cervix was gripped with a clamp. In the case of severe pain in the patient or the inability to penetrate the cervical canal, collection of the material was discontinued. Immediately after the examination, patients were asked to rate the intensity of pain during the procedure numerically on the numerical rating scale (NRS), where 0 is no pain at all and 10 is the worst pain imaginable. There were no complications in any of the patients. The collected endometrial sample was preserved in a solution of 10% neutral, buffered formalin at room temperature, and then transferred to the CMUJ Clinical and Experimental Pathology Department for fixation in paraffin blocks.

On the same day, a 5 ml venous blood sample on EDTA was collected from each patient. The blood was centrifuged for 15 minutes at 3000 rpm, and the serum was sent to the Department of Clinical Biochemistry of the Jagiellonian University Medical College for the determination of IL-18 and histamine levels.

Immunohistochemistry Tissue material was fixed in formaldehyde for 24 hours. Then it was dehydrated in 70% ethanol solution and then embedded in paraffin. Tissues were sectioned 4 µm thick and mounted on silanized slides. The sections were divided into three equal sets. Paraffin preparations were dewaxed (3 xylene exchanges at room temperature; the first exchange - 10 minutes, the second and third exchange after 15 minutes) and rehydrated (3 alcohol exchanges at room temperature, 5 minutes each). Then the preparations were incubated at room temperature for 10 min. in a 3% H2O2 solution to block endogenous peroxidase. Slides were rinsed in distilled water and incubated with TBS for 5 minutes. Then the slides were unmasked with citrate buffer pH 6.0 in a water bath at 97 ° C. After the preparations were unmasked, the Ultra Vision Protein Block preparation (Thermo Scientific) was applied for 5 min. at room temperature in a humid chamber. Then the appropriate antibody was applied and incubated at room temperature in a humid chamber for a specified time (Table 1). The first set of sections was incubated with IL-18 reactive rabbit polyclonal antibodies (Recombinant IL18 (Tyr37 ~ Asp193), Cloud-Clone Corp., 0.33 mg / ml Cat. No. PAA064HU01) at a dilution of 1:00 for 60 min. The second set was incubated with histamine reactive rabbit polyclonal antibodies (Recombinant human histamine (Met1 ~ Ile163), Cloud-Clone Corp., 0.35mg / ml, catalog no. PAA927Ge01) at a dilution of 1: 100 for 30 min. The third set was incubated with rabbit polyclonal antibodies (Recombinant human GLUT4 (Met1 ~ Ile163) Cloud-Clone Corp., catalog no. PAC023HU01) at a dilution of 1:50 for 30 min. Excess antibody was washed with TBS buffer and Post antibody blocking for Bright Vision plus (BrightVision + Goat anti-mouse / rabbit HRP - ImmunoLogic kit) was applied. We incubate in a humid chamber at room temperature for 20 minutes.

Excess reagent was washed off with TBS buffer and a poly-HRP-GAMs / Rb IgG preparation (BrightVision + Goat anti-mouse / rabbit HRP - ImmunoLogic kit) was applied. Incubated at room temperature in a humid chamber for 30 minutes. Excess reagent was washed off with TBS buffer and DAB Quanto (Thermo Scientific) was applied. Incubated at room temperature in a humid chamber for about 5 minutes. Then, the excess reagent was rinsed with distilled water and the slides were colored with hematoxylin (Thermo Scientific). The preparations were dehydrated by carrying out a series of three changes of alcohol and xylene in increasing concentrations. Closed with a coverslip (CYTOSEAL by ThermoScientific). Expression of each cytokine was assessed semi-quantitatively as the number of positive cells per square millimeter in the analyzed sample, calculated using an image analyzer.

IL-18 and histamine in the blood Serum IL-18 measurement was performed by ELISA using human recombinant IL-18 (Human IL-18 ELISA Kit, Biorbyt, catalog no. Orb50153). Blood samples and reagents were warmed to 37 ° C and then diluted 1: 2 with the diluent using 50 µL of buffer with complete and uniform mixing. The solution was dispensed 0.1 ml per well. The microliter plate with the wells was covered with a lid and incubated at 37 ° C for 90 min. The plate was then dried, 0.1 ml of biotinylated anti-human IL-18 antibody solution was added to each well and incubated at 37 ° C for 60 min. The plate was then washed three times in 0.01 M TBS (TRIS buffered saline), each time leaving the wash buffer in the well for 1 min. The buffer was removed and the plate was dried, then 0.1 ml of prepared avidin-biotin-peroxidase (ABC) solution was added to each well and the plate was incubated at 37 ° C for 30 min. The plate was rinsed again, this time 5 times with 0.01 M TBS, and the washing buffer was left in the wells for 1-2 min each time. The buffer was removed and the plate was dried, then 90 µl of TMB dye was added to each well and the plate was incubated at 37 ° C for 10 min. 0.1 ml of TMB contrast dye solution was added to each well and the absorbance was immediately measured at 450 nm. Serum histamine levels were measured by ELISA using the Histamin ELISA Immundiagnostik reagent, catalog number K 8212. The washing buffer concentrate (WASHBUF B) was diluted 1:10 in pure water. Reagents were brought to room temperature. The plasma samples were mixed with the derivatization reagent. The derivatized sample was then incubated on a horizontal shaker together with a peroxidase labeled polyclonal histamine antibody on a histamine derivative coated ELISA plate for 1 hour at room temperature. Then the contents of the wells were washed 5 times with 250 µl of the washing buffer. After the last step, residual buffer was removed with tissue paper. Then 100 μl of substrate (SUB) was pipetted into each well, incubated for 15 minutes at room temperature, protected from light. 100 µl of the contrast dye solution was added to each well. The absorbance was measured immediately at 450 nm. The results are expressed in picograms per milliliter.

Statistical analysis. Statistical analysis was performed using the Statistica program (StatSoft 13.3). The Shapiro-Wilk normality test of the examined variables and the presented frequency charts showed that the distribution of the variables was not normal. The non-parametric Wald-Wolfowitz and U Mann-Whitney tests were used to compare the study group with the control group. The significance test of the correlation coefficient was based on the statistics for the Student's t-distribution.

ELIGIBILITY:
Study group

Inclusion criteria:

* primary infertility (unsuccessfully trying to become pregnant for more than a year)
* regular menstruation

Exclusion criteria:

* female homronal therapy
* established male factor of infertility
* tubal factor
* endometriosis
* inflammation in the pelvic area - currently and in the history
* hormonal background of infertility
* obesity
* insulin resistance
* status post at least one miscarriage
* chronic autoimmune diseases.

Control group

Inclusion criteria:

* naturally conceived offspring up to three years of age
* regular menstruation

Exclusion criteria were:

* status post surgery on the uterus, including curettage of the uterine cavity
* endometriosis
* pelvic inflammation - present and in the history
* at least one miscarriage
* obesity
* insulin resistance
* chronic autoimmune diseases
* breastfeeding.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study group consisted of 58 women diagnosed with primary infertility, and a control group consisted of 8 patients with naturally conceived offspring. Patients were recruited from among women hospitalized at the Gynecological Endocrinology and Gynecology Clinic, consulted at the Gynecological Endocrinology Clinic and diagnosed under the Comprehensive Reproductive Health Program
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Il-18 in the blood | July 2017- December 2020
  Level of IL-18 in the blood in women with idiopathic infertility compared to women with children
Il-18 in endometrium | July 2017- December 2020
  Level of IL18 in endometrium in women who have children compared to women with idiopathic infertility
Histamine in the blood | July 2017- December 2020
  Histamine levels in the blood of women with idiopathic infertility compared to women who had children
Histamine in endometrium | July 2017- December 2020
  Histamine levels in the receptive endometrium of women with idiopathic infertility compared to women with children
GLUT4 in endometrium | July 2017- December 2020
  GLUT4 levels in the receptive endometrium of women with idiopathic infertility compared to women with children
Endometrium vs blood levels of histamine and Il-18 | July 2017- December 2020
  Correlation between the level of IL-18 in the endometrium and its level in the blood. Correlation between the level of histamine in the endometrium and its level in the blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic Of Endocrynological Gynecology, Krakow, Malopolska, Poland

IPD SHARING:
Plan to Share IPD: No